CLINICAL TRIAL: NCT05408351
Title: The Indonesian Version of Ages and Stages Questionnaire III Accuracy Compared to Bayley Scales of Infant Development III
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Prof. Hartono Gunardi, MD, PhD, Professor, Indonesia University
Other Study IDs: 1005/UN2.F1/ETIK/PPM.00.02
Record Dates: First submitted 2022-05-25; First posted 2022-06-07 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Child Development; Child Development Disorder; Development Delay; Developmental Delay; Global Developmental Delay; Motor Delay; Speech Delay
Keywords: ASQ-3; BSID-III; child development; Indonesia; screening test; validity
MeSH Terms: conditions — Developmental Disabilities; Learning Disabilities; Psychomotor Disorders; Language Development Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to evaluate the concurrent validity information of the 24-, 30-, and 36-month Indonesian ASQ-3 with the Bayley Scales of Infant and Toddler Development 3rd Edition (BSID-III) in Indonesian children. Children living in Tanah Tinggi subdistrict, Central Jakarta, were recruited conveniently from November to December 2019. Children within the 24-, 30-, or 36-month age group were assessed for Indonesian ASQ-3 concurrently with BSID-III as the reference standard according to their age groups. Screening test accuracy was measured in sensitivity, specificity, and predictive values for both overall dan specific domains.

ELIGIBILITY:
Inclusion Criteria:

* Parents with children aged 23 - 38 months
* Parents who finished at least elementary school

Exclusion Criteria:

* Parents with communication difficulties
* Parents who could not speak Indonesian language

Ages: 23 Months to 38 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Parents with children aged 23-38 months living in Central Jakarta.
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Child development | Day 1
  Measured once with Indonesian Ages and Stages-3 questionnaire (cross sectional study) with scores ranging between 0 to 60 per domain. Higher score means better development.
Child development | Day 1
  Measured once with Bayley Scales Infant Development-III with scores ranging between 40 to 160 per domain. Higher score means better development.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanah Tinggi subdistrict community health centers, Jakarta Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided